CLINICAL TRIAL: NCT06801353
Title: A Cohort Study on Biomarkers to Predict the Efficacy of Biologics for Chronic Rhinosinusitis with Nasal Polyps
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR-Biological treatment of NP
Record Dates: First submitted 2025-01-13; First posted 2025-01-30 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-12

CONDITIONS: Chronic Rhinosinusitis with Nasal Polyps (CRSwNP); Biological Therapy; Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- therapy group (Experimental): Stapokibart subcutaneously every two weeks plus mometasone furoate nasal spray 200 μg once daily
  Interventions: Biological: Stapokibart; Drug: Mometasone Furoate Nasal Spray (MFNS)

INTERVENTIONS:
Biological: Stapokibart — Stapokibart subcutaneously every two weeks
Drug: Mometasone Furoate Nasal Spray (MFNS) — mometasone furoate nasal spray 200 μg once daily

SUMMARY:
Recently, several biologic therapies have become available for treating chronic rhinosinusitis with nasal polyps (CRSwNP). However, not every patient responds to these treatments. This clinical trial aims to develop a non-invasive predictive model to help determine how effective IL-4Rα targeted monoclonal antibody therapy will be for individuals with CRSwNP.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old.
2. With bilateral chronic rhinosinusitis with nasal polyposis.
3. Nasal Polyp Score ≥4 (minimum score of 2 per nasal cavity) at baseline.
4. Nasal congestion score ≥2 at baseline.
5. Patients who have received systemic corticosteroids (SCS) treatment within 2 years before screening, and/or have contraindications or intolerance to SCS treatment, and/or received surgical for nasal polyps more than 6 months before screening.
6. Have been using intranasal corticosteroids (INCS) at a stable dose for at least 4 weeks before screening.
7. Symptoms of nasal obstruction and additional symptoms such as loss of smell or rhinorrhea should be present for at least 4 weeks before screening.
8. Good adherence.

Exclusion Criteria:

1. Not enough washing out period for prior biological therapy (within 10 weeks or 5 half-lives [whichever is longer] before baseline).
2. Use of systemic immunosuppressants for inflammatory diseases or autoimmune diseases within 8 weeks or 5 half-lives before baseline (whichever is longer).
3. Initiation of leukotriene receptor antagonist treatment, oral glucocorticoid treatment, or traditional Chinese medicine treatment for chronic rhinosinusitis within 4 weeks before baseline.
4. Subjects who have undergone surgery that changed the nasal structure and cannot be evaluated for Nasal Polyp Score.
5. Participants with a forced expiratory volume in 1 second (FEV1) ≤50% of predicted normal during screening/run-in period.
6. Hypersensitivity to MFNS or anti-IL-4R monoclonal antibodies or stapokibart components.
7. Concomitant with other poorly controlled serious diseases or recurrent chronic diseases.
8. Women who are pregnant, breastfeeding, or planning either during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Nasal Polyps Score (NPS) | week 16
  NPS score ranges from 0-8 (sum of 0-4 for each nasal), higher score means a worse outcome.
Nasal Congestion Score (NCS) | week 16
  Change from baseline in the Nasal Congestion Score (NCS) at week 16. NCS score range from 0 to 3, with higher score means worse nasal symptom.

SECONDARY OUTCOMES:
Nasal Polyp Score (NPS) | Week 2，4，8，12，20，24，28，32，36，40
  Changes from baseline in nasal polyp score (NPS) at each evaluation time point. NPS score ranges from 0-8 (sum of 0-4 for each nasal), higher score means a worse outcome.
Nasal Congestion Score (NCS) | Week 2，4，8，12，20，24，28，32，36，40
  Changes from baseline in nasal congestion score (NCS) at each evaluation time point. NCS score range from 0 to 3, with higher score means worse nasal symptom.
sino-nasal outcome test-22 (SNOT-22) | Week 2，4，8，12，20，24，28，32，36，40
  Changes from baseline in sino-nasal outcome test-22 (SNOT-22) score at each evaluation time point. The SNOT-22 score is the sum of the scores of 22 items, ranging from 0 to 110 (higher scores indicate worse outcomes).
nasal total symptom score (TSS) | Week 2，4，8，12，20，24，28，32，36，40
  Changes from baseline in nasal total symptom score (TSS) at each evaluation timepoint. The evaluation content of TSS includes three aspects: nasal congestion, loss of smell and running nose. Each aspect has a score of 0-3 with a total score of 0-9. The higher score indicates the more severe overall symptom.
Asthma Control Questionnaire (ACQ-6) | Week 2，4，8，12，20，24，28，32，36，40
  Changes from baseline in Asthma Control Questionnaire (ACQ-6) at each evaluation timepoint for participants with asthma. The ACQ-6 is a questionnaire used to evaluate the degree of asthma control. Each question is scored from 0 to 6 according to its severity. The higher the score, the less satisfactory symptom control is.
Lund-Mackay CT score | week 16
  Change from baseline in Lund-Mackay CT score evaluated by sinus computed tomography (CT) at each evaluation timepoint. The total Lund-Mackay score ranges from 0 to 24 points. The six parts of the nasal sinuses on both sides are evaluated separately. The higher the score, the more severe the CRS condition.
Pulmonary function test | week 16
  Change from baseline in forced expiratory volume in 1 second (FEV1) at each evaluation timepoint for participants with asthma.
Change of NPS | Week 2，4，8，12，16
  Proportion of participants with ≥1 point improvement from baseline in NPS at each evaluation timepoint. Proportion of participants with ≥2 point improvement from baseline in NPS at each evaluation timepoint.
Change of NCS | Week 2，4，8，12，16
  Proportion of participants with ≥1 point improvement from baseline in NCS at each evaluation timepoint. Proportion of participants with ≥2 point improvement from baseline in NCS at each evaluation timepoint.
Pharmacodynamics | Week 4，8，12，16，20，24，28，32，36，40
  Change from baseline in serum biomarker level (eosinophil level).
Pharmacodynamics | week 16
  Change from baseline of eosinophil level in nasal polyps biospy tissue.
The change of biomarkers | Week 8，16，24，32，40
  Changes from baseline of expression levels of biomarker in nasal brush exfoliated cells, nasal secretions and nasal microbes.
Pulmonary function test | week 16
  Change from baseline in forced vital capacity (FVC) at each evaluation timepoint for participants with asthma.
Pulmonary function test | week 16
  Change from baseline in mean flow with forced expiratory volume of 25% ~ 75% vital capacity (FEF25 ~ 75%) at each evaluation timepoint for participants with asthma.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No